CLINICAL TRIAL: NCT01434407
Title: Crossover Meal Study Investigating Effects of Advanced Glycation Endproducts on Satiety and Inflammation
Brief Title: Effects of Advanced Glycation Endproducts on Satiety and Inflammation
Acronym: AGE-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government)
Responsible Party: Principal Investigator, AAstrup, Dr Med Sci, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: M200
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Type 2 Diabetes; Insulin Resistance; Cardiovascular Disease
Keywords: Advanced glycation endproducts; Satiety; Obesity; Inflammation; Insulin resistance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low AGE meal (Experimental): Test meal prepared by boiling/steaming the food
  Interventions: Other: Dietary meal intervention
- High AGE meal (Experimental): Test meal prepared by frying/grilling the food
  Interventions: Other: Dietary meal intervention

INTERVENTIONS:
Other: Dietary meal intervention — Test meals with different AGE content made by different cooking methods

SUMMARY:
The purpose of the meal study is to investigate acute effects on satiety and inflammation of advanced glycation endproducts (AGE) in healthy overweight subjects. The AGE content of the meal is affected by food preparation methods: frying/grilling versus boiling/steaming.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 20 and 50 years old
* BMI 25-40
* Waist circumference above 88 cm for women and above 102 cm for men

Exclusion Criteria:

* Exercise training above 8 hour/week
* Smoking
* Pregnant or breast-feeding women
* Post-menstrual women
* Regular use of medicine (except contraceptive pills)
* Previous gastric bypass surgery
* Donation of blood within the last 3 months
* Involvement in other clinical trials
* Allergic to paraaminobenzoic acid

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Appetite sensation | Every 30 min up to 5 hours after test meal
  Appetite sensation measured by visual analogue scales
Plasma ghrelin | Continuous measurement up to 5 hours after test meal
Plasma GLP-1 | Continuous measurements up to 5 hours after test meal
Plasma PYY | Continuous measurements up to 5 hours after test meal
Plasma insulin | Continuous measurements up to 5 hours after test meal
Plasma glucose | Continuous measurements up to 5 hours after test meal
Urine AGE | From 24 hour before to 48 hour after test meal

SECONDARY OUTCOMES:
Plasma triglycerides | Continuous measurements up to 5 hours after test meal
Expression of genes related to AGE | Continuous measurements up to 24 hours after test meal
IL-1 beta | Continuous measurements up to 5 hours after test meal
IL-6 | Continuous measurements up to 5 hours after test meal
TNF-alpha | Continuous measurements up to 5 hours after test meal
CRP | Continuous measurements up to 5 hours after test meal
VCAM | Continuous measurements up to 5 hours after test meal
ICAM | Continuous measurements up to 5 hours after test meal
MIF | Continuous measurements up to 5 hours after test meal
Plasma AGE | Continuous measurements up to 48 hours after test meal
Urine isoprostanes | From 24 hour before to 24 hours after test meal

CONTACTS AND LOCATIONS:
Overall Officials: Susanne G Bügel, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Human Nutrition, University of Copenhagen, Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Poulsen MW, Bak MJ, Andersen JM, Monosik R, Giraudi-Futin AC, Holst JJ, Nielsen J, Lauritzen L, Larsen LH, Bugel S, Dragsted LO. Effect of dietary advanced glycation end products on postprandial appetite, inflammation, and endothelial activation in healthy overweight individuals. Eur J Nutr. 2014;53(2):661-72. doi: 10.1007/s00394-013-0574-y. Epub 2013 Aug 9. PMID 23929260